CLINICAL TRIAL: NCT02157246
Title: RHYTHM-I: Modulation of Radiotherapy According to HYpoxia: Exploiting Changes in the Tumour Microenvironment to Improve Outcome in Rectal Cancer.
Brief Title: RHYTHM-I: Investigating Hypoxia in Rectal Tumours
Acronym: RHYTHM-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OCTO_043
Record Dates: First submitted 2013-10-10; First posted 2014-06-05 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Hypoxia in Rectal Cancer
Keywords: hypoxia; rectal cancer
MeSH Terms: conditions — Hypoxia; Rectal Neoplasms | interventions — pimonidazole; Biopsy; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A, pimonidazole, no CRT (Other): Biopsy, Blood sample, F-MISO PET, pCT, functional MRI, Pimonidazole
  Interventions: Other: Pimonidazole; Other: F-MISO PET; Other: pCT; Other: Functional MRI; Procedure: Biopsy; Procedure: Blood sample
- Group B, CRT (Other): Biopsy, Blood sample, F-MISO PET, pCT, functional MRI
  Interventions: Other: F-MISO PET; Other: pCT; Other: Functional MRI; Procedure: Biopsy; Procedure: Blood sample

INTERVENTIONS:
Other: Pimonidazole
  Arms: Group A, pimonidazole, no CRT
Other: F-MISO PET
Other: pCT
Other: Functional MRI
Procedure: Biopsy
Procedure: Blood sample

SUMMARY:
A low level of oxygen in cancer cells makes them less likely to respond to chemotherapy and radiotherapy treatments. There is interest in using new drugs that improve the level of oxygen in tumours. Another approach would be to increase the radiotherapy dose to tumours with low oxygen levels.

Before we can do this for patients with rectal cancer, we need to develop a reliable way of identifying areas of low oxygen within the rectal tumour. This will make us able to tell which patients may be suitable for such a change in their treatment.

Traditionally, the level of oxygen in tumours is measured by inserting a needle into the tumour and measuring it directly. This is not possible in rectal cancer. This study has been designed to identify the best alternative method. We would like to do a blood test, take samples of cancer tissue and some detailed scans (18F-fluoromisonidazole (F-MISO) positron emission tomography, perfusion computed tomography, functional magnetic resonance imaging). The results of these tests will be compared to decide which gives us the most comprehensive and reliable information.

Patients in Group A go straight to surgery. By looking for markers of low oxygen levels on the tumour that has been removed, we will be able to find out which of the study tests performed before the tumour was removed is the best. By repeating the scans we will be able to see how reliable they are and how much they change on a day to day basis. We think that tumours that still have low levels of oxygen after 8 to 10 doses of radiotherapy are the least likely to respond to treatment.

Group B will have scans before radiotherapy treatment and after 8 to 10 doses of radiotherapy to see if we can identify the patients that have persistent low levels of oxygen.

ELIGIBILITY:
Inclusion Criteria (Group A):

1. T2-3 N0 histologically proven adenocarcinoma of the rectum (if the MDT has an index of suspicion of malignancy high enough to proceed to surgical resection despite repeatedly non-diagnostic biopsies, the patient should be considered eligible).
2. The tumour on MRI and/or CT measures at least 2 cm by 2 cm.
3. MRI confirmation that the circumferential resection margin is not involved or threatened
4. Agreement from the local multi-disciplinary team (MDT) that the tumour is operable and does not require pre-operative CRT.
5. The patient is medically fit for operative resection of the tumour.
6. Male or female, Age at least 18 years.
7. ECOG performance score of 0-2 and be capable of co-operating with protocol.
8. Written (signed and dated) informed consent.
9. Haematological and biochemical indices within the ranges shown below:

   1. Haemoglobin (Hb) ≥12.0 g/dL
   2. Platelet count ≥ 100 x 109/L
   3. PT 10-14 seconds
   4. Renal function:

Serum Creatinine <120 mmol/L OR Calculated GFR >50 ml/min

Inclusion Criteria (Group B):

1. Histologically confirmed invasive adenocarcinoma of the rectum
2. Pelvic MRI defined disease:

   a. Mesorectal fascia (MRF) involved or breached i. Includes involvement of adjacent organ b. Mesorectal fascia threatened (tumour ≤ 1mm from MRF). This includes i. Primary tumour ≤ 1mm from MRF ii. Extramural vascular invasion ≤ 1mm from MRF iii. Tumour deposit with irregular border and mixed signal intensity ≤ 1mm from MRF c. Low tumours at/below the level of the levators where: i. Tumour ≤ 1mm from levator on two imaging planes ii. Tumour through full thickness of muscularis propria or beyond at level of puborectalis sling or below iii. Tumour involving the intersphincteric plane iv. Tumour involving the external anal sphincter
3. Patient is considered likely to be fit for surgical resection following CRT
4. Patient has been considered to be medically fit to receive CRT by their treating oncologist
5. Male or female, Age at least 18 years.
6. ECOG performance score of 0-2.
7. The patient is willing and able to give informed consent and to comply with the protocol for the duration of the study.
8. Haematological and biochemical indices within the ranges shown below:

   1. Haemoglobin (Hb) ≥12.0 g/dL
   2. Absolute neutrophil count ≥1.5 x 10^9/L
   3. Platelet count ≥ 100 x 109/L
   4. PT 10-14 seconds
   5. Renal function:

Serum Creatinine <120 mmol/L OR Calculated GFR >50 ml/min

Exclusion Criteria (Group A):

1. Unequivocal evidence of metastatic disease. Patients with equivocal lesions will be determined as eligible on consensus of the MDT.
2. Previous pelvic radiotherapy.
3. Pregnant or breast-feeding women, or women of childbearing potential unless effective methods of contraception are used.
4. Treatment with any other investigational agent, or participation in another interventional clinical trial within 28 days prior to enrolment.
5. Currently taking anti-coagulants
6. Patients who for any reason are unable to undergo MRI and/or CT scans as per local guidelines e.g. if they are fitted with a pacemaker, have metal fragments in or around the eye, cannot tolerate the scan for any reason or are allergic to contrast agents.
7. Patients who are known to be serologically positive for Hepatitis B, Hepatitis C or HIV.

Exclusion Criteria (Group B):

1. Previous pelvic radiotherapy (including brachytherapy)
2. Unequivocal evidence of metastatic disease. Patients with equivocal lesions will be determined as eligible on consensus of the MDT.
3. Pregnant or breast-feeding women, or women of childbearing potential unless effective methods of contraception are used.
4. Currently taking anti-coagulants
5. Gastrointestinal disorder which would interfere with oral therapy and its bioavailability
6. Treatment with any other investigational agent, or participation in another clinical trial within 28 days prior to enrolment.
7. Other psychological, social or medical condition, physical examination finding or a laboratory abnormality that the Investigator considers would make the patient a poor trial candidate or could interfere with protocol compliance or the interpretation of trial results.
8. Patients who for any reason are unable to undergo MRI and/or CT scans as per local guidelines e.g. they are fitted with a pacemaker, have metal fragments in or around the eye, cannot tolerate the scan for any reason or are allergic to contrast agents.
9. Patients who are known to be serologically positive for Hepatitis B, Hepatitis C or HIV.

Exclusion Criteria (Optional supplemental oxygen breathing Groups A and B):

1. Ongoing supplemental oxygen as part of clinical care
2. Known lung disease with carbon dioxide retention
3. Chronic obstructive airways disease with known or at risk of hypercapnia
4. Most recent available arterial blood gas (ABG) from the current hospital admission demonstrates hypoxia or hypercapnia on room air.
5. Any patient not felt to be suitable for supplemental oxygen as considered by an appropriately trained clinician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Group A FMISO-PET derived hypoxic volumes | At surgery
  Validation of FMISO-PET as a measure of hypoxia in rectal cancer.
  FMISO-PET derived hypoxic volumes will be compared to reconstructed volumes from the immunohistochemistry of PIMO, CAIX and HIF on whole mount histology of the resected tumour.
  The spatial distribution of FMISO uptake on PET images will be compared with PIMO, CAIX and HIF immunohistochemistry distributions in the resected tumour.
Group B Percentage change in FMISO-PET SUVmax and uptake volume | Day -7 to -2 and day 10-12
  Quantifying the percentage change in FMISO SUVmax and uptake volume between the two FMISO-PET scans after 8-10 fractions of CRT.

SECONDARY OUTCOMES:
Hypoxia gene microarray read outs from biopsies | Day -7 to -2 (Group A & B) and day 10-12 (Group B)
  Group A: To assess if F-MISO PET defined hypoxia correlates with hypoxia metagene expression.
  Group B: To assess if baseline measures of hypoxia and the presence of tumour hypoxia after 8-10 fractions of CRT correlate with radiological/pathological response.
FMISO-PET SUVmax | Day -7 to -2 (Group A & B) and 10-12 (Group B only)
  Group A: Assess inter-individual variability in FMISO uptake and intra-individual reproducibility of FMISO-PET in rectal cancer.
  Group B: Determine correlation of baseline and day 10-12 FMISO-PET SUVmax with radiological/pathological response, immunohistochemical and genetic markers of hypoxia and other factors affecting response to radiotherapy following CRT.
pCT derived blood flow parameters | Day -7 to -2 (Group A & B) and day 10-12 (Group B)
  Group A: Assess inter-individual variability in pCT derived blood flow parameters and intra-individual reproducibility of pCT in rectal cancer. Assessment of the utility of pCT derived AIF in the processing of dynamic FMISO-PET scans.
  Group B: Quantitative changes in pCT derived blood flow parameters after 8-10 fractions of CRT.
Comparison of changes in T1/T2* MRI | Prior to Day -7 (Group A), Day -21 to Day -1 (Group B), Day 10-12 (Group B)
  Group A: Comparison of changes in T1/T2* MRI before and after supplemental oxygen breathing.
  Group B: Changes in native T1/T2* MRI from baseline and before and after supplemental oxygen breathing.

OTHER OUTCOMES:
Blood sample | Day -7 to -2 and day 10-12
  Blood samples will be taken at each imaging time point for investigational work to identify potential circulating hypoxia biomarkers.
F-MISO PET hypoxic volumes and pCT images | Prior to Day -7 (Group A)
  Comparison of F-MISO PET hypoxic volumes with fractal analysis of pCT images.
Radiotherapy planning feasibility study | Day 10-12 (Group B)
  Radiotherapy planning feasibility study to determine if it is feasible to change the radiotherapy dose distribution or total dose in response to functional imaging after 8-10 fractions of radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Maughan, Principal Investigator — University of Oxford
Locations (1):
- Oxford University Hospitals NHS Trust, Oxford, United Kingdom